CLINICAL TRIAL: NCT06004765
Title: A Prospective Single-center Study on the Efficacy and Safety of Lenalidomide Combined With Azacitidine vs Azacitidine in the Treatment of MDS-RS
Brief Title: Efficacy and Safety of Lenalidomide Combined With Azacitidine vs Azacitidine in the Treatment of MDS-RS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Len+Aza-MDS-RS
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lenalidomide and sequential azacitidine (Experimental): Lenalidomide (10mg/d *21 days, 28 days for 1 course), at least 2 courses. If effective, continue to use lenalidomide until ineffective or intolerant. Patients receive azacitidine (75mg/m2/d*5 days, 28 days for 1 course). Until progression or intolerance. At least 2 sessions of treatment are needed.
  Interventions: Drug: Lenalidomide; Drug: Azacitidine
- azacitidine (Experimental): Azacitidine (75mg/m2/d*5 days, 28 days for 1 course) for at least 4 courses
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Lenalidomide — 10mg/d *21 days, 28 days for 1 course
  Arms: lenalidomide and sequential azacitidine
Drug: Azacitidine — 75mg/m2/d*5 days, 28 days for 1 course

SUMMARY:
At present, the main therapies for myelodysplastic syndromes with ring sideroblasts (MDS-RS) are red blood cell and platelet transfusion, erythropoietin (EPO), androgen, and iron chelation therapy. Lenalidomide is an immunomodulator with multiple mechanisms, including direct targeting of MDS clones, immunomodulation, erythropoiesis restoration, and angiogenesis inhibition. A Phase III, randomized, placebo-controlled trial of oral azacitidine (AZA) in lower-risk MDS reported higher rates of hemoglobin and platelet hematological improvement in patients with AZA monotherapy. Therefore, this study intended to investigate the efficacy and safety of lenalidomide and sequential AZA in the treatment of refractory MDS-RS versus azacitidine monotherapy.

DETAILED DESCRIPTION:
Myelodysplastic neoplasms (MDS) are heterogeneous clonal disorders of stem cells that result in peripheral blood cytopenia and ineffective hematopoiesis, with the potential risk of the development of acute myeloid leukemia (AML). Most patients with myelodysplastic syndromes with ring sideroblasts (MDS-RS) are stratified into lower-risk groups by the revised International Prognostic Scoring System (IPSS). At present, the main therapies for MDS-RS are red blood cell and platelet transfusion, erythropoietin (EPO), androgen, and iron chelation therapy. Lenalidomide is an immunomodulator with multiple mechanisms, including direct targeting of MDS clones, immunomodulation, erythropoiesis restoration, and angiogenesis inhibition. Hypomethylating agents (HMA) like azacytidine (AZA) and decitabine (DEC), have been shown to improve survival or delay disease progression in high-risk MDS. A Phase III, randomized, placebo-controlled trial of oral AZA in lower-risk MDS reported higher rates of hemoglobin and platelet hematological improvement in patients with AZA monotherapy (24.3% vs 6.5%). Therefore, this study intended to investigate the efficacy and safety of lenalidomide and sequential azacitidine in the treatment of refractory MDS-RS versus azacitidine monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Patients with a definite diagnosis of MDS-RS and stratified as lower-risk according to IPSS-R.
3. After at least 3 months of rhEPO treatment, with hemoglobin<90g/L, absolute neutrophil count≥1.0× 109 /L, and platelet≥30× 109 /L
4. Unconditional hematopoietic stem cell transplantation
5. Adequate hepatic functions with alanine transaminase (ALT)/aspartate. transaminase (AST) levels within 2 times of the normal upper limit and total bilirubin levels within 2 times of the normal upper limit.

5. No active infection; Not pregnant or breastfeeding 6. ECOG≦2 with an expected life span of more than 6 months 7. Documented patient consent.

Exclusion Criteria:

1. Proliferative (white blood cell count ≥12× 109 /L) chronic myelomonocytic leukemia.
2. Complicated with active or uncontrolled infections.
3. Complicated with other malignancies.
4. Creatinine/transaminase ≥ 2 normal upper limit.
5. Complicated with myelofibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 3, 6 months
  Proportion of patients achieved complete response, partial response, and hematological improvement.
complete response rate | 3, 6 months
  Proportion of patients achieved complete response.

SECONDARY OUTCOMES:
relapse free survival (RFS) | 3, 6, 12, 24 months
  Relapse free survival will be calculated from the date of response to the date of first recorded relapse or death from any cause.
Overall survival (OS) | 3, 6, 12, 24 months
  OS is calculated for all patients from the date of initial registration to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Eisenmann KM, Dykema KJ, Matheson SF, Kent NF, DeWard AD, West RA, Tibes R, Furge KA, Alberts AS. 5q- myelodysplastic syndromes: chromosome 5q genes direct a tumor-suppression network sensing actin dynamics. Oncogene. 2009 Oct 1;28(39):3429-41. doi: 10.1038/onc.2009.207. Epub 2009 Jul 13. PMID 19597464
- [Background] Kotla V, Goel S, Nischal S, Heuck C, Vivek K, Das B, Verma A. Mechanism of action of lenalidomide in hematological malignancies. J Hematol Oncol. 2009 Aug 12;2:36. doi: 10.1186/1756-8722-2-36. PMID 19674465
- [Background] Quach H, Ritchie D, Stewart AK, Neeson P, Harrison S, Smyth MJ, Prince HM. Mechanism of action of immunomodulatory drugs (IMiDS) in multiple myeloma. Leukemia. 2010 Jan;24(1):22-32. doi: 10.1038/leu.2009.236. Epub 2009 Nov 12. PMID 19907437
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Fenaux P, Giagounidis A, Selleslag D, Beyne-Rauzy O, Mufti G, Mittelman M, Muus P, Te Boekhorst P, Sanz G, Del Canizo C, Guerci-Bresler A, Nilsson L, Platzbecker U, Lubbert M, Quesnel B, Cazzola M, Ganser A, Bowen D, Schlegelberger B, Aul C, Knight R, Francis J, Fu T, Hellstrom-Lindberg E; MDS-004 Lenalidomide del5q Study Group. A randomized phase 3 study of lenalidomide versus placebo in RBC transfusion-dependent patients with Low-/Intermediate-1-risk myelodysplastic syndromes with del5q. Blood. 2011 Oct 6;118(14):3765-76. doi: 10.1182/blood-2011-01-330126. Epub 2011 Jul 13. PMID 21753188
- [Background] Santini V, Almeida A, Giagounidis A, Gropper S, Jonasova A, Vey N, Mufti GJ, Buckstein R, Mittelman M, Platzbecker U, Shpilberg O, Ram R, Del Canizo C, Gattermann N, Ozawa K, Risueno A, MacBeth KJ, Zhong J, Seguy F, Hoenekopp A, Beach CL, Fenaux P. Randomized Phase III Study of Lenalidomide Versus Placebo in RBC Transfusion-Dependent Patients With Lower-Risk Non-del(5q) Myelodysplastic Syndromes and Ineligible for or Refractory to Erythropoiesis-Stimulating Agents. J Clin Oncol. 2016 Sep 1;34(25):2988-96. doi: 10.1200/JCO.2015.66.0118. Epub 2016 Jun 27. PMID 27354480
- [Background] Garcia-Manero G, Santini V, Almeida A, Platzbecker U, Jonasova A, Silverman LR, Falantes J, Reda G, Buccisano F, Fenaux P, Buckstein R, Diez Campelo M, Larsen S, Valcarcel D, Vyas P, Giai V, Oliva EN, Shortt J, Niederwieser D, Mittelman M, Fianchi L, La Torre I, Zhong J, Laille E, Lopes de Menezes D, Skikne B, Beach CL, Giagounidis A. Phase III, Randomized, Placebo-Controlled Trial of CC-486 (Oral Azacitidine) in Patients With Lower-Risk Myelodysplastic Syndromes. J Clin Oncol. 2021 May 1;39(13):1426-1436. doi: 10.1200/JCO.20.02619. Epub 2021 Mar 25. PMID 33764805
- [Background] Silverman LR, Demakos EP, Peterson BL, Kornblith AB, Holland JC, Odchimar-Reissig R, Stone RM, Nelson D, Powell BL, DeCastro CM, Ellerton J, Larson RA, Schiffer CA, Holland JF. Randomized controlled trial of azacitidine in patients with the myelodysplastic syndrome: a study of the cancer and leukemia group B. J Clin Oncol. 2002 May 15;20(10):2429-40. doi: 10.1200/JCO.2002.04.117. PMID 12011120
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Kantarjian H, Issa JP, Rosenfeld CS, Bennett JM, Albitar M, DiPersio J, Klimek V, Slack J, de Castro C, Ravandi F, Helmer R 3rd, Shen L, Nimer SD, Leavitt R, Raza A, Saba H. Decitabine improves patient outcomes in myelodysplastic syndromes: results of a phase III randomized study. Cancer. 2006 Apr 15;106(8):1794-803. doi: 10.1002/cncr.21792. PMID 16532500